CLINICAL TRIAL: NCT03959540
Title: A Multinational, Multicentre, Prospective Non-interventional Study to Assess Safety and Effectiveness of Opicapone Plus Standard of Care in Elderly Patients With Parkinson's Disease
Brief Title: Safety and Effectiveness of Opicapone Plus Standard of Care in Elderly Patients With Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: BIA-91067-402
Record Dates: First submitted 2019-04-23; First posted 2019-05-22 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-10

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — opicapone; Levodopa; Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Standard of care (including L-DOPA) + starting opicapone
  Interventions: Drug: Opicapone; Drug: Levodopa (L-DOPA) + Standard care
- Cohort 2: Standard of care (including L-DOPA)
  Interventions: Drug: Levodopa (L-DOPA) + Standard care

INTERVENTIONS:
Drug: Opicapone — Capsules, oral use - 50 mg Use of opicapone is only driven by the physician's decision.
  Other Names: Ongentys
  Groups: Cohort 1
Drug: Levodopa (L-DOPA) + Standard care — Levodopa (immediate- or controlled-release) + Standard care. Use of Levodopa and standard of care are only driven by the physician's decision.

SUMMARY:
The purpose of this study is to describe the safety and efficacy of opicapone plus standard of care in elderly patients with PD in the real-world setting

DETAILED DESCRIPTION:
This will be a multinational, multicentre, prospective non-interventional study in elderly patients with PD. Approximately 100 patients with PD will be recruited by specialists from approximately 37 sites in European countries. The total enrolment period will be one year, and each patient will be followed for up to one year after enrolment.

PD patients with end-of-dose motor fluctuations suitable for additional treatment optimization will be included in the study and split into 2 cohorts:

* Cohort 1: 50 patients; standard of care (including L-DOPA) + starting opicapone
* Cohort 2: 50 patients; standard of care (including L-DOPA Data will be collected at baseline (date of enrolment), 1 month, 3 months, 6 months, 9 months, and 12 months after enrolment.

This non-interventional study does not recommend the use of any specific treatments. Use of opicapone and of standard of care are only driven by the physician's decision.

ELIGIBILITY:
Inclusion Criteria:

* Patient or legally acceptable representative willing and able to provide informed consent as mandated by local regulation
* Patient with clinical diagnosis of idiopathic PD (excluding non-idiopathic PD: atypical Parkinsonism, secondary [acquired or symptomatic] Parkinsonism, Parkinson-plus syndrome)
* Patient with age >=75 years at enrolment
* Patient with end-of-dose motor fluctuations suitable for additional treatment optimization

Exclusion Criteria:

* Patient concurrently participating in any clinical trial
* Patient who used tolcapone or opicapone previously
* For the patient who starts opicapone: concomitant treatment with entacapone or tolcapone is not allowed
* Patient with any contraindications to Ongentys use
* Patient with any concomitant medical condition that could interfere with study assessments

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study plans to recruit approximately 100 elderly PD patients from neurology clinics
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2020-04-28 (Actual); Primary Completion 2021-05-11 (Actual); Study Completion 2021-05-11 (Actual)

PRIMARY OUTCOMES:
Percentage of patients having at least one Adverse Event (AE) | through study completion, an average of 1 year
  All AEs reporting

SECONDARY OUTCOMES:
Clinical Global Impression of Improvement (CGI-I) | at Follow-up visit at 1, 3, 6, 9, 12 months
  hange of score from baseline at each follow-up visit (from 0=good health to 100=poor health).
Parkinson Disease Questionnaire (PDQ-8) | at baseline, Follow-up visit at 6,12 months
  hange of score from baseline at each follow-up visit (from 0=good health to 100=poor health).
Unified Parkinson's Disease Rating Scale (UPDRS) | at baseline, Follow-up visit at 6,12 months
  change from baseline at each follow-up visit for each of the 4 sections and for the total score (from 0=no disability to 199=total disability).
Montreal Cognitive Assessment (MoCA) | at baseline, Follow-up visit at 6,12 months
  change from baseline at each follow-up visit (30-point test; score >26 is normal).
Patients' Global Impressions of Change (PGI-C) | at Follow-up visit at 1, 3, 6, 9, 12 months
  Percentage of patients for each item at each follow-up visit (from 1=very much improved since the initiation of treatment to 7=very much worse since the initiation of treatment).

CONTACTS AND LOCATIONS:
Locations (1):
- Norfolk&Norwich University Hospitals, Norwich, Norfolk, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided